CLINICAL TRIAL: NCT01481363
Title: A Feasibility Study of a Psychosocial Intervention - The Talking Sense Communication Programme for Dementia Family Carers
Brief Title: The Talking Sense Communication Programme for Dementia Carers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Portsmouth (Other)
Collaborators: Solent NHS Trust (Other Government); The Sir Halley Stewart Trust (Unknown)
Responsible Party: Principal Investigator, Mr COLIN BARNES, Principal Speech and Language Therapist and PhD student, School of Health Sciences, University of Portsmouth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOP3203201
Record Dates: First submitted 2011-11-22; First posted 2011-11-29 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Dementia
Keywords: dementia; communication; carers; caregivers; psychosocial support systems; education
MeSH Terms: conditions — Dementia; Communication | interventions — Psychosocial Intervention; Therapeutics; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment as usual (Active Comparator): Half of participants recruited will be randomly assigned to the control group to receive treatment as usual. This is will be based on a single one hour consultation which will include communication advice and information.
  Interventions: Behavioral: Treatment as usual - communication information and advice
- The Talking Sense treatment (Experimental): Half of carer participants recruited will be randomly assigned to receive the Talking Sense treatment. This will be conducted one to one and individualised over 3 sessions and no more than 4.5 hours during no more than 8 weeks.
  Interventions: Behavioral: The Talking Sense manual

INTERVENTIONS:
Behavioral: The Talking Sense manual — Talking Sense is a recently written therapy manual for professionals to use with carers of people with dementia. It is intended to be used one to one with carers and is individualisable according to their relatives degree of communication difficulty or the extent to which the carer experiences difficulty with communication. The approach addresses the carers knowledge, skills, thinking and behaviour in a series of interdependent steps. In this study it will be delivered to carers during 3 home visits and up to a total of 4.5 hours.
  Other Names: Psychosocial intervention
  Arms: The Talking Sense treatment
Behavioral: Treatment as usual - communication information and advice — Carers will receive the existing model of support provided by the speech and language therapy service. This is based on a one hour visit during which questions will be answered and specific advice given. No leaflets or manual will be used.
  Arms: Treatment as usual

SUMMARY:
Do family carers of people with dementia benefit from communication therapy and training? This study will only involve carers of people with dementia. Nearly all people with dementia will experience some difficulty communicating. Family carers of people with dementia have described communication and associated behaviour difficulties as one of the hardest to cope with.

This is a PhD study. The student/investigator has previously produced a detailed manual of approaches for supporting relatives of people with dementia who are experiencing communication difficulties. Previously published communication guides by other authors do not present research evidence.

Carers will be recruited to this study from the local NHS older person's mental health service overseen by their relative's psychiatrist. Only family carers will be included. Recruits will be randomly assigned to a treatment group or a control group. People in the control group will receive treatment as usual. The carers will be seen at home or at an NHS site if they prefer. The investigator and carer will work through the contents of the manual together. The manual is designed to consider their knowledge, thinking, skills and behaviour. The treatment will take no more than 4.5 hours over a period of up to 12 weeks.

Carers will be asked to complete questionnaires before and after the treatment. As well as background information, these questionnaires will look for any significant effects of the treatment on carers' anxiety and depression, carers' quality of life, carers' belief in their ability to care, communication difficulties experienced and the carers perceptions of their relatives communication competence.

A sample of 15 carers will also be interviewed by a third party interviewer who will be an existing speech and language therapy employee of Solent NHS Trust (see attached job description and person specification). The interviews will ask more specifically about their thoughts, feelings and opinions of this intervention and their experience in addressing communication difficulties.

DETAILED DESCRIPTION:
This is a feasibility study that intends to recruit 60 family carers over a period of up to 4 years. Carers will remain in the study for up to 12 weeks. They will be randomly assigned to a Talking Sense communication intervention and a treatment as usual control group of equal size. Quantitative and qualitative outcomes will be measured. Measures will include carer anxiety and depression, carer quality of life, carer general self efficacy and communication specific self efficacy as well as the carers rating of their relative's communication competence.

The null hypothesis for this study is that receiving the Talking Sense communication intervention would have no effect on carer reported depression, carer quality of life, carer's perception of their ability to cope with communication difficulties, carer reported experience of communication difficulties and carer reported person with dementia's communication competence. The alternative hypothesis suggests that one or more of these outcomes would be significantly greater for the treatment group in comparison to the control group.

This selection of outcome measures was identified by comparison with other treatment studies and in keeping with a theoretical framework for carer intervention studies described in a key text by Professor Richard Schulz, a prominent author in this field. Other longer term measures such as time to institutionalisation would be valuable though considered outside the remit of this study which is measuring short term effect only. If this feasibility study leads to a larger study, the longitudinal or wearing off of treatment effect would also be important to measure.

The ideal control group for this study would be carers receiving no treatment though this would be unethical. Comparison to another form of treatment e.g. a leaflet has been used in other studies though this introduces additional variables to account for. In this case treatment as usual is considered to be the most appropriate form of control condition.

Carers will be invited to participate in this study by a nurse or psychiatrist from the older person's mental health service. They will be asked if they wish to take a leaflet which broadly explains the purpose of the study and if their contact details can be passed to the chief investigator. All referrals will be approved by one of four overseeing psychiatrists.

If in agreement, the carer will be telephoned by the chief investigator. Some carers may be excluded if they do not meet the study criteria though still offered communication therapy outside of the study if required.

During this telephone contact, the chief investigator will provide a summary of the research study and answer any initial questions. If carers remain interested in participation, the chief investigator will arrange to visit them at home or on an NHS site. Carers will be sent a copy of the participant information sheet to read prior to this meeting.

At this first meeting, the carer will be given a copy of the participant information sheet which will be read to them as much as required. They will be supported in understanding this where necessary. If they are keen to participate, they will be invited to sign a consent form. They will be offered time for consideration and a return visit/meeting if required.

After the carer has signed a consent form they will be provided with a set of questionnaires to complete. Questionnaires will include a service receipt inventory and carer background information. The form and process of completing these questionnaires will be explained to them. They will then be asked to complete these questionnaires when alone. The chief investigator will arrange to collect these questionnaires.

Carers will be randomly assigned to the treatment or control group using a list of randomly generated numbers by a third party colleague employee of Solent NHS Trust.

Carers will be informed of their group assignment when the pre-treatment questionnaire packs are collected.

Carers assigned to the treatment group will be asked about arranging future appointments. They will then be sent a letter explaining what happens next including dates of agreed appointments and when to expect delivery of the post treatment questionnaires. All carers will be offered a telephone reminder to complete questionnaires if required.

Carers in both groups will continue to receive any support already planned from members of the older person's mental health service. Carers in the control group will also receive communication advice from the investigator in keeping with a model of treatment as usual. Carers in both groups will complete a service receipt inventory in their post intervention set of questionnaires.

Carers in both groups will be advised of when to expect delivery and collection of a second post-intervention set of questionnaires. These will be collected.

The referrer and over-seeing psychiatrist will be informed of the carer's decision to participate and assignment to treatment or control group.

Carers will be seen on 3 occasions for a maximum total time of 4.5 hours. All interventions will be provided by the chief investigator.

Carers will be encouraged to be seen alone. Therapy sessions will be offered in their home or at an NHS site.

Carers will be shown the Talking Sense manual and given an overview of the 9 steps that it covers: knowledge, insight, thoughts and feelings, the environment, the person, how to be as the carer, reminders and encouraging conversation, communication and activities and challenging behaviours.

All treatment session will be audio recorded. Analysis of these recordings will be used to measure the treatment provider's adherence as well as time spent on and most popular topics of discussion. Carers will also be invited to make notes.

During the first session carers will be encouraged to grade their relative's degree of communication difficulty using the grading scale incorporated into the Talking Sense programme.

The investigator will also use display resources adapted from the Talking Sense manual to explain specific issues.

For the second and third session the carers will be encouraged to select topics to discuss, thoughts to consider and strategies to rehearse from the Talking Sense programme. Suitability of topics will be guided by the grade of communication difficulty they previously selected. There are five grades: very early, early, moderate, advanced and severe. For example, the validation approach to communication in dementia is only suitable for people with moderate, advanced or severe communication difficulties in dementia.

Within one week of the final treatment session, all treatment group carers will be sent a 1-2 page printed individualised summary of the topics and issues identified and discussed.

The study period will be 10 to 12 weeks for each carer. For those receiving the intervention there will be at least a two week gap between receiving the summary document after the last intervention session and completing the post intervention questionnaires and interview.

Between weeks 10 and 12, a purposive sample of approximately 15 carers from the intervention group will be invited to participate in an interview. These will be conducted by a single independent interviewer who will be an existing Speech and Language Therapy department employee of Solent NHS Trust. This person will have been trained by the chief investigator in using a semi-structured interview protocol. Carers will be asked to participate in an interview, at a location of their choice (as above) lasting no longer than 60 minutes.

These interviews will be recorded and transcribed. The investigator will use a grounded hermeneutic approach of analysis with constant comparison leading to the development of themes and meta-themes. Consent to participate in the interview will be agreed with all participants at the start of the study until all interviews are completed.

At the end of their participation, all participants will be sent a thank you letter. Carers will also be able to request further advice and support if required.

ELIGIBILITY:
Inclusion Criteria:

Carers will be included in this study if they are:

* Spouses, co-habiting partners or children of the person with dementia in communication contact with their relative with dementia for more than two hours weekly.
* Caring for a relative with a diagnosis of Alzheimer's disease, vascular dementia or lewy body dementia.
* Reporting "existing difficulties with communication"
* Demonstrating capacity to understand and consent to participation for the duration of the study
* Considered suitable with particular attention to the carers mental wellbeing, by the overseeing or referring psychiatrist, for participating within this study.
* Only receiving interventions within the parameters of treatment as usual as defined below.
* Caring for a person with dementia with a recent score of between 21 and 27 out of 30 on the M.M.S.E. test (Folstein et al, 1975).

  * Carers demonstrating signs of anxiety and depression will not be excluded, due to its high prevalence, but will be screened as suitable for participation by the referring psychiatrist.
  * Although the Talking Sense manual is suitable for the widest range of communication difficulties in dementia, this study will limit its use to a cohort or people within the range of mild dementia as defined in the NICE clinical guidelines (2007). Using a more homogenous group of caregivers should improve generalisability of results. See also answer to question 6-2.
  * Treatment as usual will include medical, psychological and social treatments provided by health and social services including speech and language therapy for carers and people with dementia and informed by a modelling exercise of local services which is a separate objective of this Ph.D. study.
  * Carers considered to be receiving greater than standard treatment e.g. more than once weekly or other treatments focusing specifically on communication and behaviour or incorporating CBT will be excluded from participation in this study though will still be eligible for existing speech and language therapy services. It is expected that very few carers will be receiving greater than standard treatments.

Exclusion Criteria:

Carers will be excluded from participation if they:

* Have not been approved for participation by an overseeing psychiatrist
* Are caring for someone with a primary communication impairment associated with fronto-temporal dementia, Parkinson's disease or stroke as it is expected their presentation and experience will be significantly different.
* Carers who have already received any significant form of individualised communication therapy e.g. with speech and language therapy or occupational therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Hospital anxiety and depression scale (HADS) (Zigmund and Snaith, 1983) | At ten weeks
  A carer self completed measure of anxiety and depression

SECONDARY OUTCOMES:
Change from baseline in The Communication Competence Scale (Weimann et al, 1977) | At ten weeks
  A carer self completed questinonaire rating the carers' perception of their relatives communication competence.
Change from baseline in The adult carer quality of life questionnaire (Elwick et al, 2010) | At ten weeks
  A recently published scale developed specifically for carers. This is self completed by carers to judge their own quality of life.
Change from baseline in The general self efficacy scale (Schwarzer and Jerusalem, 1995) with modifications to identify communication specific self efficacy | At ten weeks
  The general self efficacy scale is a published scale which will be completed alone carers. An additional scale has been developed to identify communication specfiic self-efficacy as no published scale was availalble This has been based on communication issues identified by carers during the development of the Talking Sense trial and has undergone an evaluation of face and content validity.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Markham, Ph.D., Study Director — University of Portsmouth
Locations (1):
- Speech and Language Therapy Department, Solent NHS Trust, St James Hospital,, Portsmouth, Hamsphire, United Kingdom